CLINICAL TRIAL: NCT02818361
Title: Topical Tripterygium Wilfordii Gel for Treatment in Patients With Moderate Activity Rheumatoid Arthritis
Brief Title: Topical Tripterygium Wilfordii Gel for Moderate Activity Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Chief, Rheumatology Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z161100001816046
Record Dates: First submitted 2016-06-15; First posted 2016-06-29 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Tripterygium wilfordii Hook F; double-blinded; randomized controlled trial; Tripterygium; Administration; Topical
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- topical TwHF gel group (Experimental): Topical TwHF gel recipe composes Tripterygium wilfordii Hook F, Mangxiao (Mirabilite), Chuanxiong (Rhizoma Ligustici), Ruxiang (Olibanum), Moyao (M yrrh) (prescription proportion is 4:4:2:2:1).Each gel is 20 gram(g). TwHF gel is applied for 1st to 5th metacarpophalangeal joints, 1st to 5th proximal interphalangeal joints, wrists, knees and ankles 20g for 1 hour, once per day from week 0 through week 4 and 10g for 1 hour, once per day from week 5 through week 8.
  Interventions: Drug: Topical tripterygium gel
- placebo group (Placebo Comparator): Placebo recipe composes viscous agent which matches by the sucrose. The usage and dosage of topical TwHF and placebo are the same.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Topical tripterygium gel
  Arms: topical TwHF gel group
Drug: Placebo gel
  Arms: placebo group

SUMMARY:
Tripterygium wilfordii Hook F (TwHF), a traditional Chinese herb, is widely used in China for treating Rheumatoid Arthritis (RA), but limited only for elderly RA patients because of its reproductive system toxicity. The investigators are inspired by Chinese external therapy, an immemorial therapy for thousands of years, and take its advantage to make TwHF topically in order to get an effective and safe treatment for active RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of rheumatoid arthritis, as defined by the American Rheumatism Association 1987 Revised Criteria.
* Documented diagnosis of damp-heat syndrome according to Traditional Chinese Medicine.
* Patients, men and women, must age from 18 to 65 years old.
* Patients must have moderately active RA based on the criteria of the DAS-28 score from 3.2 to 5.1.
* If patients are receiving Disease-modifying anti-rheumatic drugs (DMARDs), then the doses should have been kept stable for at least 12 weeks.
* If patients are receiving non-steroidal anti-inflammatory drugs (NSAIDs) or orally Chinese herbal medicine, then the doses should have been kept stable for at least 4 weeks.

Exclusion Criteria:

* Skin allergies or broken skin;
* Taking TwHF agents, glucocorticoids and biological agents;
* Female patients who are pregnant, breast-feeding or planed to be pregnant;
* Subjects suffering serious hyperlipidemia, hyperglycemia, diabetes mellitus, cardiovascular diseases, gastrointestinal problems or liver and renal failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Twenty percent improvement in the American College of Rheumatology criteria | Week 8.
  a patient must have 20% or greater improvement in both tender and swollen joints (28 tender and 28 swollen joints were assessed) and 20% or greater improvement in 3 or more of the following: the physician's or patient's assessment of global health status, the patient's assessment of pain on a visual analogue scale, the patient's assessment of function using a modified version of the Health Assessment Questionnaire (HAQ), and the erythrocyte sedimentation rate (ESR) or serum C-reactive protein (CRP) level.
Twenty percent improvement in the American College of Rheumatology criteria | Week 4.

SECONDARY OUTCOMES:
Fifty percent improvement in the American College of Rheumatology criteria | Week 4 and week 8.
  a patient must have 50% or greater improvement in both tender and swollen joints (28 tender and 28 swollen joints were assessed) and 50% or greater improvement in 3 or more of the following: the physician's or patient's assessment of global health status, the patient's assessment of pain on a visual analogue scale, the patient's assessment of function using a modified version of the HAQ), and the ESR or CRP level.
The changes of the 28-joint count Disease Activity Score (DAS28) | Week 4 and week 8.
The changes of Visual Analogue Scale (VAS) pain score | Week 1, 2, 3, 4, 5, 6, 7, and 8.
The change of knee synovitis classification as assessed by musculoskeletal ultrasound (MSUS) | Week 2, 4, and 8.
  Synovitis classification is specific as follows: 0 level, no doppler signal; level 1: three independent point or 2 successive or 1 and 2 in independent dot doppler signal; level 2: doppler signal < 50% of the synovial membrane area; level 3 doppler signal is the synovium in > 50% of the area.
The change of knee synovial hyperplasia classification as assessed by MSUS | Week 2, 4, and 8.
  Synovial hyperplasia classification is specific as follows: 0 level, no synovial hyperplasia; level 1: synovial hyperplasia of mild, not more than bone surface high attachment; level 2: synovial hyperplasia more than bone surface high wire, but not more than the backbone; level 3: synovial hyperplasia more than bone surface peak wires, and extends along the backbone of the side.
The change of knee articular cavity effusion as assessed by MSUS | Week 2, 4, and 8.
  Articular cavity effusion adopts binary evaluation, namely: 0: normal, 1: abnormal.
The change of knee bone erosion classification as assessed by MSUS | Week 2, 4, and 8.
  Bone erosion classification adopts binary evaluation, namely: 0: normal, 1: abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Jiang, MD. PhD., Principal Investigator — Rheumatology Department
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Q, Tang XP, Chen XC, Xiao H, Liu P, Jiao J. Will Chinese external therapy with compound Tripterygium wilfordii hook F gel safely control disease activity in patients with rheumatoid arthritis: design of a double-blinded randomized controlled trial. BMC Complement Altern Med. 2017 Sep 5;17(1):444. doi: 10.1186/s12906-017-1957-z. PMID 28870177